CLINICAL TRIAL: NCT00482872
Title: Familial HNSCC Syndrome and p16 Germline Mutations
Brief Title: Germline Mutations in Patients With Head and Neck Cancer and a Family History of Cancer
Status: Completed | Type: Observational
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: CDR0000546713; P30CA068485 (NIH); VU-VICC-HN-0402; VICC-IRB-040030
Record Dates: First submitted 2007-06-04; First posted 2007-06-05 (Estimated); Last update posted 2017-03-14 (Actual); Status verified 2017-03

CONDITIONS: Head and Neck Cancer
Keywords: stage I squamous cell carcinoma of the hypopharynx; stage II squamous cell carcinoma of the hypopharynx; stage III squamous cell carcinoma of the hypopharynx; stage IV squamous cell carcinoma of the hypopharynx; recurrent squamous cell carcinoma of the hypopharynx; stage I squamous cell carcinoma of the larynx; stage II squamous cell carcinoma of the larynx; stage III squamous cell carcinoma of the larynx; stage IV squamous cell carcinoma of the larynx; recurrent squamous cell carcinoma of the larynx; stage I squamous cell carcinoma of the lip and oral cavity; stage II squamous cell carcinoma of the lip and oral cavity; stage III squamous cell carcinoma of the lip and oral cavity; stage IV squamous cell carcinoma of the lip and oral cavity; recurrent squamous cell carcinoma of the lip and oral cavity; metastatic squamous neck cancer with occult primary squamous cell carcinoma; recurrent metastatic squamous neck cancer with occult primary; untreated metastatic squamous neck cancer with occult primary; stage I squamous cell carcinoma of the nasopharynx; stage II squamous cell carcinoma of the nasopharynx; stage III squamous cell carcinoma of the nasopharynx; stage IV squamous cell carcinoma of the nasopharynx; recurrent squamous cell carcinoma of the nasopharynx; stage I squamous cell carcinoma of the oropharynx; stage II squamous cell carcinoma of the oropharynx; stage III squamous cell carcinoma of the oropharynx; stage IV squamous cell carcinoma of the oropharynx; stage I squamous cell carcinoma of the paranasal sinus and nasal cavity; stage II squamous cell carcinoma of the paranasal sinus and nasal cavity; stage III squamous cell carcinoma of the paranasal sinus and nasal cavity; stage IV squamous cell carcinoma of the paranasal sinus and nasal cavity; recurrent squamous cell carcinoma of the paranasal sinus and nasal cavity; salivary gland squamous cell carcinoma; recurrent verrucous carcinoma of the larynx; recurrent verrucous carcinoma of the oral cavity; stage I verrucous carcinoma of the larynx; stage I verrucous carcinoma of the oral cavity; stage II verrucous carcinoma of the larynx; stage II verrucous carcinoma of the oral cavity; stage III verrucous carcinoma of the larynx; stage III verrucous carcinoma of the oral cavity; stage IV verrucous carcinoma of the larynx; stage IV verrucous carcinoma of the oral cavity; recurrent squamous cell carcinoma of the oropharynx
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck | interventions — Gene Expression Profiling; Polymerase Chain Reaction; Amplified Fragment Length Polymorphism Analysis; Flow Cytometry

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Genetic: gene expression analysis
Genetic: mutation analysis
Genetic: polymerase chain reaction
Genetic: polymorphism analysis
Other: flow cytometry
Other: laboratory biomarker analysis

SUMMARY:
RATIONALE: Studying gene mutations in samples of DNA from patients with head and neck cancer and a family history of cancer may help doctors learn more about the development of cancer in families.

PURPOSE: This clinical trial is studying germline mutations in patients with head and neck cancer and a family history of cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Measure the incidence of p16^INK4a germline mutations in patients with squamous cell carcinoma of the head and neck and a family history of cancer.
* Determine biologic activity of identified p16^INK4a germline mutations.

OUTLINE: DNA specimens are collected for genetic and mutation analysis and examined by PCR and flow cytometry. The activity of cells with p16 mutations is determined by cell cycle arrest functional assay.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of squamous cell carcinoma (SCC) of the head and neck
* Must have ≥ 1 first-degree relative with any of the following cancers:

  * Non-small cell lung cancer
  * Melanoma
  * Pancreatic cancer
  * SCC of the head and neck
  * Lymphoma (controls)

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* Not specified

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2004-03 (Actual); Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Incidence of INK4a-p16 germline mutations
Biologic activity of identified INK4a-p16 germline mutations

CONTACTS AND LOCATIONS:
Overall Officials: Wendell G. Yarbrough, MD, FACS, Study Chair — Vanderbilt-Ingram Cancer Center
Locations (3):
- United States (3):
  - Vanderbilt-Ingram Cancer Center - Cool Springs, Nashville, Tennessee
  - Vanderbilt-Ingram Cancer Center at Franklin, Nashville, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee